CLINICAL TRIAL: NCT06398587
Title: An Open-Label, Phase II Trial to Assess Efficacy and Safety of Onvansertib in Combination With Gemcitabine and Nab-Paclitaxel in Patients With Previously Untreated, Locally-Advanced or Unresectable Pancreatic Adenocarcinoma
Brief Title: Onvansertib in Combination With Gemcitabine and Nab-paclitaxel for the Treatment of Patients With Locally-advanced, Unresectable, or Metastatic Pancreatic Ductal Adenocarcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrawal
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Charles D Lopez, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00026545; NCI-2024-02588 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00026545 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Locally Advanced Pancreatic Ductal Adenocarcinoma; Metastatic Pancreatic Ductal Adenocarcinoma; Stage II Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Unresectable Pancreatic Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — onvansertib; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; Magnetic Resonance Spectroscopy; Specimen Handling

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (onvansertib, GnP) (Experimental): Patients receive onvansertib PO QD on days 1-5, 8-12, and 15-19 and gemcitabine IV and nab-paclitaxel IV on days 1, 8, and 15. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo electrocardiography at baseline, as well as blood sample collection, tumor biopsy, CT, MRI, and/or PET throughout the trial.
  Interventions: Drug: Onvansertib; Drug: Gemcitabine; Drug: Nab-paclitaxel; Procedure: Electrocardiography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Biospecimen Collection; Procedure: Computed Tomography
- Group 2 (onvansertib monotherapy lead-in, GnP) (Experimental): Patients receive onvansertib PO QD on days 1-10. Patients then receive onvansertib, gemcitabine, and nab-paclitaxel as in Group 1. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo electrocardiography at baseline, as well as blood sample collection, tumor biopsy, CT, MRI, and/or PET throughout the trial.
  Interventions: Drug: Onvansertib; Drug: Gemcitabine; Drug: Nab-paclitaxel; Procedure: Electrocardiography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Biospecimen Collection; Procedure: Computed Tomography

INTERVENTIONS:
Drug: Onvansertib — Given PO
  Other Names: NMS-1286937; PCM 075; PCM-075; PLK-1 Inhibitor PCM-075; PLK1 Inhibitor PCM-075; Polo-like Kinase 1 Inhibitor NMS-1286937; Polo-like Kinase 1 Inhibitor PCM-075
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Paclitaxel Nanoparticle Albumin-bound; Paclitaxel Protein-Bound; Protein-bound Paclitaxel
Procedure: Electrocardiography — Undergo electrocardiography
  Other Names: ECG; EKG
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Specimen Collection
Procedure: Biospecimen Collection — Undergo tumor biopsy
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography

SUMMARY:
This phase II trial studies how well onvansertib in combination with gemcitabine and nab-paclitaxel works in treating patients with pancreatic ductal carcinoma (PDAC) that has spread to nearby tissue or lymph nodes (locally advanced), that cannot be removed by surgery (unresectable), or that has spread from where it first started (primary site) to other places in the body (metastatic). Onvansertib is a small chemical molecule that binds and stops the function of of PLK1 in tumor cells. By attacking the PLK1 protein, onvansertib is thought to reduce tumor cells ability to replicate and grow; causing them to die. Chemotherapy drugs, such as gemcitabine and nab-paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy with onvansertib may kill more tumor cells in patients with locally-advanced, unresectable, or metastatic pancreatic ductal carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess preliminary response to treatment with onvansertib and gemcitabine and nab-paclitaxel (GnP).

SECONDARY OBJECTIVES:

I. To assess the safety of onvansertib in combination with GnP. II. To assess the rate of disease control following treatment with onvansertib and GnP in patients with PDAC.

III. To estimate the duration of response (DOR). IV. To estimate the time to disease progression. V. To estimate the progression-free survival associated with onvansertib and GnP.

VI. To estimate the overall survival associated with onvansertib and GnP.

EXPLORATORY OBJECTIVE:

I. To evaluate therapy induced changes in the tumor and tumor ecosystem.

OUTLINE: This is a safety lead-in study of onvansertib in combination with GnP, followed by a phase II study. Patients are assigned to 1 of 2 groups.

GROUP 1: Patients receive onvansertib orally (PO) once daily (QD) on days 1-5, 8-12, and 15-19 and gemcitabine intravenously (IV) and nab-paclitaxel IV on days 1, 8, and 15. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo electrocardiography at baseline, as well as blood sample collection, tumor biopsy, computed tomography (CT), magnetic resonance imaging (MRI), and/or positron emission tomography (PET) throughout the trial.

GROUP 2: Patients receive onvansertib PO QD on days 1-10. Patients then receive onvansertib, gemcitabine, and nab-paclitaxel as in Group 1. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo electrocardiography at baseline, as well as blood sample collection, tumor biopsy, CT, MRI, and/or PET throughout the trial.

Upon completion of the study treatment, patients are followed up at 30 days and then every 3 months for up to 12 months from date of last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Must provide written informed consent before any study-specific procedures or interventions are performed
* Must be ≥ 18 years old at the time of informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Histologically or cytologically-proven adenocarcinoma of the exocrine pancreas with locally advanced or metastatic disease
* Must not have received prior radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease. Prior palliative radiotherapy of metastases for alleviation of pain is permitted provided that irradiated metastases are not target lesions
* Patient must be eligible to receive GnP regimen for the treatment of their PDAC in accordance with institutional standards
* Must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1
* Must have at least one disease lesion that is amenable to biopsy procedures performed per institutional standards

  * Group 1 participant must agree to undergo two (2) research biopsies
  * Group 2 participants must agree to undergo three (3) research biopsies
* Hemoglobin ≥ 8.0 g/dL
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (> 1500 per mm^3)
* Platelet count ≥ 100 x 10^9/L (> 100,000 per mm^3);
* Creatinine ≤ 1.5 x upper limit of normal (ULN), or measured or calculated creatinine clearance > 50 mL/min/1.73 m^2 (per Cockcroft-Gault equation)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT): ≤ 3 x ULN, or ≤ 5 x ULN in presence of liver metastases
* Participants of childbearing potential (POCBP) must agree to abstain from sexual intercourse or use effective non-hormonal methods of contraception starting with the first dose of study therapy through 90 days from the last dose of study intervention
* POCBP may participate provided they have a negative serum pregnancy test at screening and a negative serum OR urine pregnancy test within 7 days of starting treatment
* Sperm-producing participants must agree to abstain from sexual intercourse or use effective contraception starting with the first dose through 1 month after last dose of study intervention

Exclusion Criteria:

* Concomitant use of other anti-cancer therapy (chemotherapy, immunotherapy, hormonal therapy (hormone replacement therapy is acceptable), radiotherapy (except for palliative), biological therapy or other novel agent) or live virus and live bacterial vaccines while receiving study medication
* Prior treatment with a PLK1 inhibitor
* Known severe hypersensitivity to onvansertib, gemcitabine, or nab-paclitaxel, or to any excipient of these medicinal products, or history of allergic reactions attributed to compounds of similar chemical or biologic composition
* Major surgery within 6 weeks prior to enrollment
* Uncontrolled intercurrent illness including symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, and myocardial infarction within 3 months of initiating study intervention
* QT interval with Fridericia's correction (QTcF) > 470 milliseconds

  * The QTcF should be calculated based on a mean of triplicate electrocardiogram (ECGs). In the case of potentially correctible causes of QT prolongation (e.g., medications, hypokalemia), the triplicate ECG may be repeated once during Screening and that result may be used to determine eligibility
  * Use of concomitant medications known to increase QTc or risk of Torsades. These drugs should only be used if there are no other alternatives and only with appropriate monitoring (i.e., electrocardiograms)
  * Presence of risk factors for torsade de pointes, including family history of Long QT Syndrome or uncorrected hypokalemia
* Known dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally
* Use of strong CYP3A4 or UGT1A1 inhibitors or strong CYP3A4 inducers. Individuals currently receiving these agents who are able to switch to alternate therapy are still eligible for participation

  * CYP3A4 or UGT1A1 inhibitors should be stopped at least one week prior to the first dose of onvansertib
  * CYP3A4 inducers should be stopped at least two weeks prior to the first dose of onvansertib
* Psychiatric illness/social situations that would limit compliance with study requirements
* Any concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, infection, hypertension, etc.)
* Participant is pregnant or breastfeeding, or expecting to conceive or sire children within the projected duration of the trial, starting with the screening visit through 90 days after the last dose of trial treatment
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-05-04 (Estimated); Study Completion 2027-06-07 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 3 months after last dose of study intervention
  Defined as the percentage of participants that achieve a best overall response of complete response (CR) or partial response (PR) (per Response Evaluation Criteria in Solid Tumors version [v]1.1 criteria). Using the Group 1 efficacy analysis set, an estimate of ORR will be reported with 95% exact confidence interval (CI).

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (AEs) and serious AEs | Up to 30 days after last dose of study intervention
  Using safety analysis set, the incidence of having treatment-emergent AEs and SAEs per Common Terminology Criteria for Adverse Events (CTCAE) 5.0 will be determined for participants that received at least one dose of onvansertib. The 95% CI will be reported with the point estimate of toxicity rate.
Disease control rate (DCR) | Up to 1 year after last dose of study intervention
  Defined as percentage of participants who have achieved CR, PR, or stable disease (SD) (per RECIST v1.1 criteria) for at least 16 weeks from initiating study treatment. Using the Group 1 efficacy analysis set, the estimate of DCR will be reported with 95% exact CI.
Duration of response (DOR) | From the date of first response (CR, PR, or SD ≥ 16 weeks [per RECIST v1.1 criteria]) to date of disease progression or death, whichever occurs first, assessed up to 1 year after last dose of study intervention
  Using the Group 1 efficacy analysis set, DOR will characterized using the Kaplan-Meier (KM) method at specific timepoints (e.g., 3, 6, 9, 12, and 24 months; median DOR), along with corresponding 95% CI.
Time to progression (TTP) | From the start of study intervention until first objectively documented date of disease progression, assessed up to 1 year after last dose of study intervention
  Using the Group 1 efficacy analysis set, the time to progression distribution will be characterized using the KM method. KM curves of TTP will be presented. Median TTP, quartiles and TTP rate after specific time points (e.g., 3, 6, 9, 12, and 24 months; median TTP) will be estimated from the survival curves. All these parameter estimates will be reported together with their 95% CIs.
Progression-free survival (PFS) | From first dose of study drug to the first date of objectively documented disease progression, or death by any cause, assessed up to 1 year from last dose of study intervention
  The estimated distribution of the PFS will be plotted using KM curves and reported with median survival and 95% CIs if available.
Overall survival (OS) | From date of first dose of study drug to the date of death by any cause, assessed up to 1 year after last dose of study intervention
  The estimated distribution of the OS will be plotted using KM curves and reported with median survival and 95% CIs if available.

CONTACTS AND LOCATIONS:
Overall Officials: Charles D Lopez, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States